CLINICAL TRIAL: NCT06934811
Title: Evaluating the Impact of Ciprofol on Oxygenator Performance in Patients Undergoing Extracorporeal Membrane Oxygenation: A Single-Center Randomized Controlled Trial (CIP-OXY Study)
Brief Title: Ciprofol's Impact on Oxygenator Function in Extracorporeal Membrane Oxygenation (ECMO) Patients
Acronym: CIP-OXY
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Principal Investigator, First Affiliated Hospital of Wannan Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202507
Record Dates: First submitted 2025-03-29; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: ECMO Treatment; ARDS (Acute Respiratory Distress Syndrome); ECMO and Acute MI; Respiratory Failure Patients Treated With ECMO; Shock, Cardiogenic
Keywords: Ciprofol; ECMO; Oxygenator function; Sedative; Randomized Controlled Trial; Midazolam; Oxygenator thrombosis
MeSH Terms: conditions — Acute Lung Injury; Shock, Cardiogenic | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ciprofol group (Experimental): Patients in this arm will receive Ciprofol, an investigational sedative, administered via continuous intravenous infusion.
  Dosing Protocol:
  Initial Dose: 0.1 mg/kg loading dose over 1-2 minutes. Maintenance Dose: 0.05-0.3 mg/kg/h, adjusted hourly based on the Richmond Agitation-Sedation Scale (RASS) score (target range: -3 to 0).
  Combined Analgesia:
  All patients will concurrently receive remifentanil (0.05-0.3 μg/kg/min) for pain control.
  Monitoring & Adjustments:
  Sedation depth assessed every 30 minutes using RASS and ( Critical-Care Pain Observation Tool) CPOT scores.
  Dose adjustments made to avoid hypotension (Mean Arterial Pressure) MAP < 65 mmHg or oversedation.
  Triglyceride levels monitored daily to guide lipid emulsion management.
  Safety Measures:
  Rescue protocol for hypotension (e.g., vasopressors) or respiratory depression (e.g., temporary ECMO flow adjustment).
  Interventions: Drug: Ciprofol
- Midazolam group (Active Comparator): Patients in this arm will receive midazolam, a benzodiazepine sedative commonly used in ECMO patients, administered via continuous intravenous infusion.
  Dosing Protocol:
  Initial Dose: 0.05 mg/kg loading dose over 2-5 minutes. Maintenance Dose: 0.02-0.1 mg/kg/h, adjusted hourly based on the RASS score (target range: -3 to 0).
  Combined Analgesia:
  All patients will concurrently receive remifentanil (0.05-0.3 μg/kg/min) for pain control, identical to the Ciprofol group.
  Monitoring & Adjustments:
  Sedation depth assessed every 30 minutes using RASS and CPOT scores, consistent with the experimental group.
  Dose adjustments made to avoid hypotension (MAP < 65 mmHg) or oversedation. Daily monitoring of drug accumulation markers (e.g., midazolam plasma levels if available).
  Safety Measures:
  Rescue protocol for hypotension (e.g., vasopressors) or respiratory depression (e.g., ventilator support escalation).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ciprofol — Continuous intravenous infusion (0.05-0.3 mg/kg/h), adjusted hourly based on the RASS score (target range: -3 to 0).
  Arms: Ciprofol group
Drug: Midazolam — Continuous intravenous infusion (0.02-0.1 mg/kg/h), adjusted hourly based on the RASS score (target range: -3 to 0).
  Arms: Midazolam group

SUMMARY:
This study evaluates the safety and effectiveness of Ciprofol, a new sedative, in critically ill patients receiving Extracorporeal Membrane Oxygenation (ECMO), a life-support system for heart or lung failure. The investigation aims to:

Assess how Ciprofol affects the oxygenator, a critical ECMO component responsible for adding oxygen to blood.

Compare the safety of Ciprofol to midazolam, a commonly used sedative. Eligibility Criteria Adults aged 18 years or older. Patients receiving ECMO and mechanical ventilation for over 72 hours. Individuals requiring sedation for medical procedures. Study Protocol

Participants will be randomly assigned to one of two groups:

Ciprofol Group: Initial sedation dose of 0.1 mg/kg, adjusted as needed. Midazolam Group: Initial sedation dose of 0.05 mg/kg, adjusted as needed. Both groups will receive pain management with remifentanil. Sedation levels will be adjusted daily by the clinical team to ensure patient safety and comfort.

Outcome Measures Primary: Oxygenator performance (oxygen and carbon dioxide levels) on Days 3 and 7.

Secondary: Changes in blood triglyceride and clotting marker (D-dimer) levels, oxygenator lifespan before replacement, and safety outcomes such as low blood pressure, respiratory issues, or allergic reactions.

Significance ECMO patients often require prolonged sedation, but current sedatives like midazolam may contribute to oxygenator damage. Ciprofol's potential for faster recovery and fewer side effects could improve sedation practices and device longevity in this high-risk population.

ELIGIBILITY:
1. Inclusion Criteria:

   * Receiving ECMO therapy with an anticipated duration exceeding 72 hours;
   * Requiring invasive mechanical ventilation;
   * Requiring sedation and analgesia treatment.
2. Exclusion Criteria:

   * BMI >45 kg/m²;
   * Age <18 years;
   * Severe hepatic (Child-Pugh Class C) or renal failure (eGFR <15 mL/min/1.73m²);
   * History of severe psychiatric disorders;
   * Pregnancy;
   * Refusal to sign informed consent;
   * Contraindications to midazolam and propofol use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite Oxygenator Dysfunction | At Day 3 and Day 7 of ECMO support
  Definition: Meeting ≥2 of the following:
  Post-oxygenator PaO₂/FiO₂ <200 mmHg ΔTransmembrane pressure (ΔdP) ≥20% from baseline or Transmembrane pressure (TMP)>50 mmHg from baseline CO₂ clearance <20% [(Pre-MLCO₂ - Post-MLCO₂)/Pre-MLCO₂] at gas flow ≥10 L/min

SECONDARY OUTCOMES:
Oxygenator Transmembrane Pressure (TMP) Gradients | Daily from Day 1 to Day 7
  Transmembrane pressure (TMP) will be assessed using continuous inline pressure monitoring via the ECMO circuit's integrated pressure sensors (e.g., pre- and post-oxygenator pressure transducers). TMP is calculated as:
  TMP (mmHg) = Post-oxygenator Pressure - Pre-oxygenator Pressure
Post-oxygenator Oxygenation Index (PaO₂/FiO₂ Ratio) | Daily from Day 1 to Day 7
  The post-oxygenator PaO₂/FiO₂ ratio will be measured daily to evaluate oxygenator efficiency. A value <200 mmHg indicates impaired oxygenation capacity.
Oxygenator Lifespan | Through ECMO weaning or Day 30, whichever comes first
  Definition: Time (hours) from ECMO initiation to oxygenator replacement. Replacement Criteria: Meeting ≥2 composite dysfunction criteria.
Lipid Profile Changes | At 24 hours, 72 hours, and Day 7
  Measure: Serum triglycerides (TG)
Plasma D-dimer Concentration (μg/mL) | At 24 hours, 72 hours, and Day 7 post-ECMO initiation.
  Description: Absolute plasma D-dimer levels measured as a biomarker of hypercoagulability and thromboembolic risk.
  Threshold: >5 μg/mL (defined as high thrombotic risk per International Society on Thrombosis and Haemostasis [ISTH] guidelines).
Incidence of delirium | At 24h post-sedation discontinuation
ECMO Pump Head Malfunction | During ECMO support (up to 30 days)
  Definition: Occurrence of any of the following:
  Pump head rupture (visible crack or leak) Pump head thrombosis (ultrasound-confirmed thrombus within the pump housing) Mechanical failure (unplanned pump stoppage requiring emergency intervention)
Thromboembolic Events | From ECMO initiation until 48 hours after decannulation
  Definition: Radiologically confirmed:
  Arterial embolism: Cerebral or limb artery occlusion (CT angiography/ultrasound) Venous thrombosis: Lower extremity DVT or pulmonary embolism (CT pulmonary angiography/Doppler) Intracardiac thrombus: Echocardiographic or CT evidence
  Grading:
  Major: Life-threatening or requiring intervention (e.g., thrombectomy) Minor: Asymptomatic or managed medically
ECMO Weaning Success | Through study completion (Day 30)
  Definition: Successful decannulation without re-initiation of ECMO within 24 hours.
7-day mortality rate | At Day 7
  All-cause death rate at Day 7 post-ECMO initiation.
28-day mortality rate | At Day 28
  All-cause death rate at Day 28 post-ECMO initiation.
ICU Length of Stay (LOS) | Through hospital discharge, up to 90 days
  Duration from ICU admission to discharge (days).
Duration of Mechanical Ventilation | From ECMO initiation to successful extubation (up to 28 days)
  Measure: Time (hours) from intubation to sustained extubation (48 hours without reintubation).

IPD SHARING:
Plan to Share IPD: No